CLINICAL TRIAL: NCT02852395
Title: A First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-48816274
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JNJ-48816274
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108090; 48816274EDI1001 (Other: Janssen-Cilag International NV); 2015-004186-89 (EudraCT Number)
Record Dates: First submitted 2016-07-11; First posted 2016-08-02 (Estimated); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 Single Dose (Experimental): Part 1 single daytime oral dose of JNJ-48816274 or placebo. Doses of JNJ-48816274 will start at 5 milligram (mg) and increase sequentially to a maximum dose of 250 mg.
  Interventions: Drug: JNJ-48816274; Drug: Placebo
- Part 2 Crossover Sleep Study (Experimental): Part 2 single nighttime oral dose of JNJ-48816274 or placebo administered during each of 3 or 4 crossover periods separated by 7-9 days. The doses of JNJ-48816274 will be selected based on data from Part 1 (not to exceed 250 mg).
  Interventions: Drug: JNJ-48816274; Drug: Placebo
- Part 3 Repeated Dose (Optional) (Experimental): Part 3 daytime oral dose of JNJ-48816274 or placebo administered once daily for 7 consecutive days. Doses will be determined based on data from Part 1, and may increase sequentially (not to exceed 250 mg/day).
  Interventions: Drug: JNJ-48816274; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-48816274 — Oral dose; dose range of 5 mg up to 250 mg
Drug: Placebo — Oral dose; appearance matched to JNJ-48816274

SUMMARY:
This is a 3-part study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of JNJ-48816274 in healthy participants after administration of single and repeated doses, and to evaluate its potential effectiveness for treating insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy as assessed by medical history and safety evaluations performed at screening
* Has a body mass index between 18 and 30 kilogram per square meter (kg/m2) and body weight not less than 50 kg
* Must be willing and able to abide by the prohibitions and restrictions of the study, including requirements for contraception
* Women must not be of childbearing potential by either being postmenapausal or permanently sterilized
* Part 2 Only: Maintains a regular sleep-wake cycle as measured by sleep diaries and a watch that measures activity
* Has a habitual (majority of days) bedtime and duration of sleep that meet the study requirements

Exclusion Criteria:

* Current or history of clinically significant medical or psychiatric illness, or recent major surgery or blood loss/donation
* Any current sleep-wake disorder, recent night shift work, or history of insomnia within the last 5 years
* Man who has a pregnant female partner
* Woman who is breastfeeding
* Is participating or has participated within the last 3 months in a study with an investigational drug or medical device
* Tests positive or has a history of human immunodeficiency virus (HIV), hepatitis B, hepatitis C, or other active liver disease
* Drug or alcohol abuse within the last 5 years, nicotine use within the last 3 months, or tests positive for alcohol, drugs of abuse, or nicotine
* Routinely consumes an excessive amount of caffeine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-08-13 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events as a Measure of Safety and Tolerability | Up to 14 days after last dose in Part 1 (approximately 5.5 weeks)
Area Under the Plasma Concentration-Time Curve From Time Zero to Time 't' (AUC[0-t]) | Days 1-2 in Part 1
Maximum Observed Plasma Concentration (Cmax) | Day 1 in Part 1
Time to Reach the Maximum Plasma Concentration (Tmax) | Day 1 in Part 1
Elimination Half Life (t1/2) | Days 1-2 in Part 1
Mean Karolinska Sleepiness Scale score | Day 1 in Part 1
  A 1-item questionnaire completed by participants to rate their degree of sleepiness on a scale of 1 to 9, ranging from 'extremely alert' (1) to 'very sleepy, great effort to keep awake, fighting sleep' (9).

SECONDARY OUTCOMES:
Mean Total Sleep Time by 8-hour overnight Polysomnography | Part 2: Days 1-2 of each of 3 or 4 crossover periods
  The sum of all minutes of sleep stages 1, 2, 3, and 4 will be assessed.
Mean Latency to Persistent Sleep by 8-hour overnight Polysomnography | Part 2: Days 1-2 of each of 3 or 4 crossover periods
  Elapsed time from the beginning of the polysomnography recording to the onset of continuous sleep will be assessed.
Mean Leeds Sleep Evaluation Questionnaire (LSEQ) Score | Part 2: Day 2 of each of 3 or 4 crossover periods
  A participant-reported 10-item visual analogue scale used to rate the quality of sleep. A 100 millimeter (mm) line used for ratings, with higher scores representing better sleep-wake characteristics.
Mean Subjective Quality of Sleep Questionnaire (SQSQ) Item Scores | Part 2: Day 2 of each of 3 or 4 crossover periods
  A participant-reported 10-item questionnaire to estimate the time to fall asleep, duration of sleep, number of awakenings, sleep quality, and feeling upon awakening.
Mean Karolinska Sleepiness Scale score | Part 2: Days 1-2 of each of 3 or 4 crossover periods; Part 3: Days 1-7
  A 1-item questionnaire completed by participants to rate their degree of sleepiness on a scale of 1 to 9, ranging from 'extremely alert' (1) to 'very sleepy, great effort to keep awake, fighting sleep' (9).
Area Under the Plasma Concentration vs. Time Curve in Subjects who are Fasted Predose vs. Those Fed a Meal | Part 1: Days 1-2
  Evaluation of the effect of food consumption on PK of JNJ-48816274.
Correlation Between Plasma Levels of JNJ-48816274 and Karolinska Sleepiness Scale Score | Day 1 of Parts 1 and 3
  Evaluation of the pharmacokinetic and pharmacodynamic relationship of JNJ-48816274 using a measure of somnolence.
Correlation Between Plasma Levels of JNJ-48816274 and Duration of Sleep as Measured by 8-hour Overnight Polysomnography | Part 2: Days 1-2 of each of 3 or 4 crossover periods
  Evaluation of the pharmacokinetic and pharmacodynamic relationship of JNJ-48816274 using a measure of sleep

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (2):
- United Kingdom (2):
  - Guildford
  - United Kingdom